CLINICAL TRIAL: NCT00409838
Title: A Phase III, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Abatacept Administered Intravenously in Korean Subjects With Active Rheumatoid Arthritis While Receiving Methotrexate
Brief Title: A Phase III Study of Abatacept in Patients With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-124
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, with inadequate response to methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abatacept and Methotrexate (Experimental)
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Placebo and Methotrexate (Placebo Comparator): (standard of care)
  Interventions: Drug: Methotrexate; Drug: Placebo
- Abatacept - Open Label (Experimental): Open-label extension phase
  Interventions: Drug: Abatacept; Drug: Methotrexate

INTERVENTIONS:
Drug: Abatacept — Intravenous (IV) solution, - weight tiered (500 mg <60 kg); (750 mg 60-100 kg); (1 gram > 100 kg), Day 1, Day 15, Day 29; every 28 days thereafter, 6 months
  Other Names: Orencia; BMS-188667
  Arms: Abatacept and Methotrexate
Drug: Methotrexate — Tablets, Oral, ≥ 15 mg, weekly, 6 months
  Arms: Abatacept and Methotrexate; Placebo and Methotrexate
Drug: Placebo — IV solution, Intravenous, D5W, Day 1, Day 15, Day 29; every 28 days thereafter, 6 months
  Arms: Placebo and Methotrexate
Drug: Abatacept — Solution, intravenous, 10 mg/kg, every 28 days
  Other Names: Orencia; BMS-188667
  Arms: Abatacept - Open Label
Drug: Methotrexate — Tablets, oral, 15 mg weekly to be adjusted according to patient condition
  Arms: Abatacept - Open Label

SUMMARY:
The purpose of the study is to demonstrate the clinical efficacy of abatacept (body-weight tiered dose approximating 10 mg/kg) compared with placebo on a background of methotrexate after 6 months (Day 169) of treatment in Korean patients with active rheumatoid arthritis and an inadequate clinical response to methotrexate

ELIGIBILITY:
Key Inclusion Criteria:

* Rheumatoid arthritis (RA) for longer than 1 year from the time of the initial diagnosis of RA
* Patients must have been taking methotrexate for at least 3 months with at least a weekly dose of 15 mg, and a stable dose for 28 days prior to treatment (Day 1)
* Methotrexate weekly dose as low as 10 mg is permitted for patients who cannot tolerate higher doses

Key Exclusion Criteria:

* Evidence (as assessed by the Investigator) of active or latent bacterial or viral infections at the time of potential enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- South Korea (5):
  - Local Institution, Seoul, Sungdong-Gu
  - Local Institution, Anyang
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Seoul

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept, 10 mg/kg: Short-term Period: Participants received a body-weight tiered dose of abatacept approximating 10 mg/kg. Study medication was administered intravenously (IV) on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141 (6-month treatment).
  Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
- Placebo: Placebo was administered IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141 (6-month treatment).
Period: Short-term Period
Arm/Group | Abatacept, 10 mg/kg | Placebo
Started | 56 (Randomized) | 57 (Randomized)
Treated (Baseline) Population | 55 | 57
Completed | 53 | 52 (Participants who received placebo in this period received abatacept in next period.)
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Never Treated | 1 | 0
Period: Long-term Extension Period
Arm/Group | Abatacept, 10 mg/kg | Placebo
Started | 105 | 0
Completed | 87 | 0
Not Completed | 18 | 0
Not completed — Adverse Event | 10 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Poor compliance/noncompliance | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept: Dosage: 500 mg to 1 g; participants randomized to the abatacept group received a body-weight tiered dose approximating 10 mg/kg. Study medication was administered intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141 (6 month treatment).
- Placebo: Study medication was administered intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141 (6 month treatment).
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 55 | 57 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.2) | 49.9 (10.6) | 48.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — One participant was randomized to the abatacept arm but never treated, and is not included in baseline characteristics.
  Participants
    Female | 47 | 49 | 96
    Male | 8 | 8 | 16
weight [Mean (Standard Deviation); unit: kilograms] | 56.5 (9.5) | 54.2 (7.5) | 55.3 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting the Criteria of the American College of Rheumatology for 20% Improvement (ACR20)
Description: The ACR 20 is based on 20% improvement (compared with baseline values) in tender and swollen joint counts and on 20% improvement in 3 of the remaining 5 core set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function) and 1 acute phase reactant value.
Time Frame: At Day 169
Population: All randomized participants who received study drug.
Measure: Number; unit: percentage of participants
Groups:
- Abatacept, 10 mg/kg: Participants received abatacept in a body-weight tiered dose approximating 10 mg/kg intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141.
- Placebo: Participants received placebo IV on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 55 | 57
percentage of participants | 65.5 | 42.1

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) ACR50 and ACR70 Response at Day 169
Description: The ACR defines ACR 50 and ACR70 response as a 50% or 70% improvement (compared with baseline values) in tender and swollen joint counts and 50% or 70% improvement in 3 of the remaining 5 core set measures (patient global assessment of pain, patient global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function) and 1 acute phase reactant value (C-reactive protein).
Time Frame: At Day 169
Population: All randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Abatacept: Participants received abatacept in a body-weight tiered dose approximating 10 mg/kg administered intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141.
- Placebo: Participants received placebo intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141.
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
Percentage of participants
  ACR 50 | 32.7 | 15.8
  ACR 70 | 14.5 | 7.0

3. Secondary Outcome: Percentage of Participants With at Least 20%, 50%, or 70% Improvement From Baseline in American College of Rheumatology (ACR) Core Components
Description: The ACR defines improvement in core components as 20%, 50%, or 70% improvement in tender and swollen joint counts and 3 of the remaining core components: patient global assessment of disease activity, physician global assessment of disease activity, patient assessment of pain, patient self-assessed disability (Health Assessment Questionnaire Disability Index [HAQ-DI]), and levels of 1 acute phase reactant (C-reactive protein levels or erythrocyte sedimentation rate.) The HAQ-DI assesses a patient's level of functional ability via 20 questions in 8 categories of functioning; scale=0 (no disability) to 3 (completely disabled); total possible score=24. The higher the score, the greater the disability.
Time Frame: From Baseline to Day 169
Population: All randomized participants who received study drug and who were evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 53 | 52
Percentage of participants
  Tender Joints ≥ 20% improvement | 81.1 | 76.9
  Tender Joints ≥ 50% improvement | 66.0 | 50.0
  Tender Joints ≥ 70% improvement | 49.1 | 23.1
  Swollen Joints ≥ 20% improvement | 92.5 | 76.9
  Swollen Joints ≥ 50% improvement | 77.4 | 57.7
  Swollen Joints ≥ 70% improvement | 60.4 | 40.4
  Patient Pain Assessment ≥ 20% improvement | 73.6 | 53.9
  Patient Pain Assessment ≥ 50% improvement | 47.2 | 23.1
  Patient Pain Assessment ≥ 70% improvement | 28.3 | 11.5
  HAQ-DI ≥ 20% improvement | 67.9 | 44.2
  HAQ-DI ≥ 50% improvement | 32.1 | 23.1
  HAQ-DI ≥ 70% improvement | 20.8 | 5.8
  Patient Global Assessment ≥ 20% improvement | 66.0 | 53.9
  Patient Global Assessment ≥ 50% improvement | 39.6 | 21.2
  Patient Global Assessment ≥ 70% improvement | 26.4 | 11.5
  Physician Global Assessment ≥ 20% improvement | 86.8 | 71.2
  Physician Global Assessment ≥ 50% improvement | 60.4 | 40.4
  Physician Global Assessment ≥ 70% improvement | 30.2 | 19.2
  C-reactive Protein ≥ 20% improvement | 83.0 | 61.5
  C-reactive Protein ≥ 50% improvement | 75.5 | 53.9
  C-reactive Protein ≥ 70% improvement | 64.2 | 28.9

4. Secondary Outcome: Change From Baseline in Disease Activity Scores (DAS) Based on C-reactive Protein (DAS 28 [CRP]) Levels or Erythrocyte Sedimentation Rate (DAS 28[ESR])
Description: Adjusted mean change from baseline. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission). CRP or ESR give estimations of DAS28 values on a group level. Change from Baseline=Postbaseline - Baseline value.
Time Frame: From Baseline to Days 169 and 1485
Population: All randomized participants who received study drug and who were evaluable.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
Units on a scale
  Day 169: DAS28 (CRP) | -2.12 (0.17) | -1.21 (0.17)
  Day 169: DAS28 (ESR) | -2.22 (0.17) | -1.15 (0.16)
  Day 1485: DAS28 (CRP) (n=31, 35) | -2.97 (0.23) | -3.13 (0.22)
  Day 1485: DAS28 (ESR) (NA) | NA (NA) — Not evaluated | NA (NA) — Not evaluated

5. Secondary Outcome: Change From Baseline to Day 169 in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: Adjusted mean change from baseline. The HAQ-DI assesses a patient's level of functional ability via 20 questions in 8 categories of functioning. Patients respond on a scale from 0 (no disability) to 3 (completely disabled); total possible score=24. Higher score indicates greater disability. Change from baseline= postbaseline - baseline value.
Time Frame: From Baseline to Day 169
Population: All randomized participants who received study drug
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
Units on a scale
  HAQ Disability Index | -0.53 (0.07) | -0.24 (0.07)
  Dressing and Grooming | -0.58 (0.09) | -0.37 (0.09)
  Arising | -0.58 (0.10) | -0.36 (0.10)
  Eating | -0.52 (0.09) | -0.13 (0.09)
  Walking | -0.54 (0.10) | -0.23 (0.10)
  Hygiene | -0.37 (0.09) | -0.21 (0.09)
  Reaching | -0.34 (0.11) | -0.11 (0.10)
  Gripping | -0.67 (0.11) | -0.36 (0.11)
  Activities | -0.56 (0.10) | -0.25 (0.10)

6. Secondary Outcome: Change From Baseline to Day 169 in Analysis of Short-Form 36 (SF-36) Health Survey Questionnaire Domains
Description: Adjusted mean change from baseline. The SF-36 is a 36-item self-administered questionnaire developed to assess health-related quality of life and comprised of 8 domains( including 4 physical and 4 mental subscales) used to derive the physical and mental component summary scores. All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from 0 to 100, with a higher score indicating better quality of life. Change from baseline=postbaseline - baseline value.
Time Frame: From Baseline to Day 169
Population: All randomized participants who received study drug and were evaluable.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 54 | 53
Units on a scale
  Physical Component Summary | 6.52 (1.05) | 2.16 (1.06)
  Mental Component Summary | 8.18 (1.37) | 4.36 (1.38)

7. Secondary Outcome: Percentage of Participants Experiencing Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs), Related SAEs and AEs, and Discontinuations Due to SAEs and AEs During the Double-Blind Period
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Throughout double-blind study period (up to Day 169); table includes data up to 56 days past double-blind period or start of the open-label period, whichever occurred first.
Population: All randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
Percentage of participants
  Deaths | 0 | 1.8
  SAEs | 3.6 | 5.3
  Related SAEs | 0 | 1.8
  Discontinued due to SAEs | 0 | 1.8
  AEs | 70.9 | 70.2
  Related AEs | 12.7 | 15.8
  Discontinued due to AEs | 0 | 1.8

8. Secondary Outcome: Abatacept Pharmacokinetic (PK) Parameters: Time to Maximum Concentration (Tmax) and Half-Life of Elimination (T-Half)
Description: Steady-state PK parameters following administration of body-weight tiered doses approximating 10 mg/kg. Tmax = the time after administration of a drug when the maximum plasma concentration is reached; when the rate of absorption equals the rate of elimination. T-Half = the biological half-life or elimination half life of a substance is the time it takes for a substance to lose half of its pharmacologic, physiologic, or radiologic activity.
Time Frame: At the end of infusion and 2 to 4 hours after the start of infusion on Day 85, at anytime between Day 92 and 96, and pre-dose on Day 113
Population: Participants with measurement at stated dose level
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
Hours
  Tmax | 1.385 (1.0607) | 1.193 (0.9956) | 1.325 (1.0351)
  T-Half | 183.583 (35.2606) | 172.451 (28.7270) | 180.078 (33.4795)

9. Secondary Outcome: Abatacept Pharmacokinetic (PK) Parameters - Maximum Concentration (Cmax)
Description: Steady-state PK parameters following administration of body-weight tiered doses approximating 10 mg/kg. Maximum Concentration (Cmax)= the maximum plasma concentration of the drug.
Time Frame: At the end of infusion and 2 to 4 hours after the start of the infusion on Day 85, at anytime between Day 92 and 96, and pre-dose on Day 113
Population: Participants with measurement at stated dose level
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
μg/mL | 241.972 (41.7191) | 312.591 (63.3026) | 264.204 (59.0589)

10. Secondary Outcome: Abatacept Pharmacokinetic (PK) Parameters - Area Under the Curve (AUC)
Description: Area Under the Plasma Concentration-Time Curve (AUC), a measure of drug absorption, in a dosing interval of 28 days from Day 85 to Day 113. Steady-state PK parameters following administration of body-weight tiered doses approximating 10 mg/kg.
Time Frame: At the end of infusion, 2 to 4 hours after the start of infusion on Day 85, anytime between Day 92 and 96, and predose on Day 113
Population: Participants with measurement at stated dose level
Measure: Mean (Standard Deviation); unit: μg.h/mL
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
μg.h/mL | 38940.063 (9731.0561) | 48283.479 (10283.2572) | 41881.508 (10743.8152)

11. Secondary Outcome: Abatacept Pharmacokinetic (PK) Parameters: Total Body Clearance (CLT)
Description: Steady-state PK parameters following administration of body-weight tiered doses approximating 10 mg/kg. Clearance is a pharmacokinetic parameter that describes how quickly drugs are eliminated, metabolized or distributed throughout the body.
Time Frame: Day 29, every 28 days until Day 141
Population: Participants with measurement at stated dose level
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
mL/h/kg | 0.269 (0.0730) | 0.240 (0.0460) | 0.260 (0.0666)

12. Secondary Outcome: Abatacept Pharmacokinetic (PK) Parameters: Volume at Steady State (VSS)
Description: The volume of distribution of drug at steady state (VSS). Steady-state PK parameters following administration of body-weight tiered doses approximating 10 mg/kg.
Time Frame: as for outcome 10
Population: Participants with measurement at stated dose level
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
L/kg | 0.064 (0.0165) | 0.055 (0.0142) | 0.061 (0.0162)

13. Secondary Outcome: Summary Statistics of Minimum Observed Serum Concentration (Cmin) for Abatacept
Description: Minimum concentration (Cmin) of Abatacept 500 mg and 750 mg at given time points
Time Frame: At the end of infusion and 2 to 4 hours after the start of the infusion on Day 85
Population: Participants with measurement at timepoint
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Abatacept 500 mg | Abatacept 750 mg | Abatacept 500 mg and 750 mg
Number analyzed (Participants) | 37 | 17 | 54
μg/mL
  Day 29 | 37.76 (10.971) | 52.19 (19.619) | 42.30 (15.611)
  Day 57 | 19.96 (11.337) | 24.42 (7.697) | 21.31 (10.504)
  Day 85 | 17.45 (7.442) | 20.83 (10.749) | 18.52 (8.661)
  Day 113 | 17.51 (6.858) | 22.06 (9.365) | 18.94 (7.936)

14. Secondary Outcome: Immunogenicity of Abatacept- Number of Participants With Reactivity Toward CTLA4-IG and CTLA4-T at Day 169
Description: Immunogenicity was determined by measuring adult subject sera for reactivity against the whole Abatacept molecule (CTLA4Ig) and CTLA4-T (CTLA4 without the Ig regions).
Time Frame: Day 169
Population: All participants who received study drug (abatacept)
Measure: Number; unit: participants
Groups:
- Abatacept + Background Methotrexate: Dosage: 500 mg to 1 g; subjects randomized to the abatacept group received a body-weight tiered dose approximating 10 mg/kg. Study medication was administered intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141 (6 month treatment).
Arm/Group | Abatacept + Background Methotrexate
Number analyzed (Participants) | 55
participants
  Reactivity toward CTLA4-T | 0
  Reactivity toward CTLA4Ig | 0

15. Secondary Outcome: Change From Baseline in Surrogate Marker Erythrocyte Sedimentation Rate (ESR) at Day 169
Description: Mean change in surrogate marker mean ESR. A surrogate marker is an indirect measurement of effectiveness. Change from Baseline = postbaseline - baseline value.
Time Frame: From Baseline to Day 169
Population: All randomized participants who received study drug. Participants with baseline and post-baseline measurements were included, not the participants who had only baseline measurements.
Measure: Mean (Standard Error); unit: mm/h
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
mm/h | -30.0 (2.86) | -4.44 (3.87)

16. Secondary Outcome: Change From Baseline in Surrogate Marker Rheumatoid Factor (RF) at Day 169
Description: Mean change in RF. A surrogate marker is an indirect measurement of effectiveness. Mean change from Baseline = postbaseline - baseline value.
Time Frame: Baseline, Day 169
Population: All Randomized and Treated Participants. The summary was based on the last observation carried forward (LOCF) procedure. Participants with baseline and post-baseline measurements were included, not the participants who had only baseline measurements.
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 55 | 57
IU/mL | -54.1 (20.52) | -12.1 (14.38)

17. Primary Outcome: Long-term Extension (LTE) (Open-Label) Period: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Related SAEs, Discontinuatons Due to SAEs, Adverse Events (AEs), Related AEs, and Discontinuations Due to AEs
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Day 169 to up to 56 days post the last dose (Day 1485) in the LTE period
Population: All participants who completed the short-term period and received at least 1 infusion of abatacept during the LTE period
Measure: Number; unit: Participants
Groups:
- All Treated: Abatacept, administered intravenously IV monthly at a fixed dose of approximately 10 mg/kg for an average of approximately 41 months in the LTE period on a background of methotrexate
Arm/Group | All Treated
Number analyzed (Participants) | 105
Participants
  Deaths | 1
  SAEs | 41
  Related SAEs | 10
  Discontinuations due to SAEs | 8
  AEs | 100
  Related AEs | 45
  Discontinuations due to AEs | 10

18. Secondary Outcome: LTE Period: Overall Number of Participants With Positive Results of Immunogenicity Samples
Description: Positive antibody titers were identified by validated enzyme-linked immunosorbent assay results. On-treatment samples were obtained during the LTE period, and posttreatment samples were following the last infusion of study medication.
Time Frame: Days 169, at 6-month intervals on-treatment, and at Days 28, 56, and 85 after the last infusion of study medication in the LTE period
Population: All participants who during the LTE period, received at least 1 infusion of abatacept and had at least 1 immunogenicity sample collected.
Measure: Number; unit: Participants
Groups:
- All Treated: Abatacept was administered intravenously monthly at a fixed dose of approximately 10 mg/kg in the LTE period on a background of methotrexate
Arm/Group | All Treated
Number analyzed (Participants) | 105
Participants
  Overall | 14
  On-treatment | 9
  Posttreatment | 11

19. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR50, and ACR70 Over Time
Description: The ACR 20, ACR50, and ACR70 are based on 20%, 50% and 70% improvement, respectively, (compared with baseline values) in tender and swollen joint counts and on 20%, 50% and 70%, respectively, improvement in 3 of the remaining 5 core set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function) and 1 acute phase reactant value.
Time Frame: Days 15 through 1569
Population: All participants who completed the ST period and received at least 1 infusion of abatacept during the LTE period. n=evaluable participants at that timepoint for that measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Abatacept, 10 mg/kg: Short-term Period: Abatacept administered IV in a body-weight tiered dose approximating 10 mg/kg. Study medication was administered on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141. LTE Period: Abatacept, administered IV monthly at a fixed dose of approximately 10 mg/kg for an average of approximately 41 months on a background of methotrexate.
- Placebo: Short-term Period: Placebo administered IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. LTE Period: Abatacept, administered IV monthly at a fixed dose of approximately 10 mg/kg for an average of approximately 41 months on a background of methotrexate.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
Percentage of participants
  Day 15 ACR20 | 13.2 [4.1 to 22.3] | 11.5 [2.9 to 20.2]
  Day 15 ACR50 | 1.9 [0.0 to 10.1] | 3.8 [0.5 to 13.2]
  Day 15 ACR70 | 0 [NA to NA] | 0 [NA to NA]
  Day 29 ACR20 | 24.5 [12.9 to 36.1] | 21.2 [10.1 to 32.3]
  Day 29 ACR50 | 1.9 [0.0 to 10.0] | 7.7 [2.1 to 18.5]
  Day 29 ACR70 | 1.9 [0.0 to 10.0] | 3.8 [0.5 to 13.2]
  Day 57 ACR20 (n=52, 52) | 51.9 [38.3 to 65.5] | 23.1 [11.6 to 34.5]
  Day 57 ACR50 (n=52, 52) | 5.8 [1.2 to 15.9] | 7.7 [2.1 to 18.5]
  Day 57 ACR70 (n=52, 52) | 1.9 [0.0 to 10.3] | 5.8 [1.2 to 15.9]
  Day 85 ACR20 | 58.5 [45.2 to 71.8] | 36.5 [23.5 to 49.6]
  Day 85 ACR50 | 17.0 [6.9 to 27.1] | 9.6 [1.6 to 17.6]
  Day 85 ACR70 | 5.7 [1.2 to 15.7] | 7.7 [2.1 to 18.5]
  Day 113 ACR20 | 64.2 [51.2 to 77.1] | 48.1 [34.5 to 61.7]
  Day 113 ACR50 | 30.2 [17.8 to 42.5] | 11.5 [2.9 to 20.2]
  Day 113 ACR70 | 3.8 [0.5 to 13.0] | 7.7 [2.1 to 18.5]
  Day 141 ACR20 | 66.0 [53.3 to 78.8] | 53.8 [40.3 to 67.4]
  Day 141 ACR50 | 30.2 [17.8 to 42.5] | 11.5 [2.9 to 20.2]
  Day 141 ACR70 | 15.1 [5.5 to 24.7] | 7.7 [2.1 to 18.5]
  Day 169 ACR20 | 67.9 [55.4 to 80.5] | 46.2 [32.6 to 59.7]
  Day 169 ACR50 | 34.0 [21.2 to 46.7] | 17.3 [7.0 to 27.6]
  Day 169 ACR70 | 15.1 [5.5 to 24.7] | 7.7 [2.1 to 18.5]
  Day 197 ACR20 (n=53, 50) | 75.5 [63.9 to 87.1] | 60.0 [46.4 to 73.6]
  Day 197 ACR50 (n=53, 51) | 45.3 [31.9 to 58.7] | 37.3 [24.0 to 50.5]
  Day 197 ACR70 (n=53, 51) | 22.6 [11.4 to 33.9] | 11.8 [2.9 to 20.6]
  Day 225 ACR20 | 75.5 [63.9 to 87.1] | 65.4 [52.5 to 78.3]
  Day 225 ACR50 | 49.1 [35.6 to 62.5] | 32.7 [19.9 to 45.4]
  Day 225 ACR70 | 22.6 [11.4 to 83.9] | 13.5 [4.2 to 22.7]
  Day 253 ACR20 (n=52, 51) | 71.2 [58.8 to 83.5] | 64.7 [51.6 to 77.8]
  Day 253 ACR50 (n=52, 51) | 44.2 [30.7 to 57.7] | 35.3 [22.2 to 48.4]
  Day 253 ACR70 (n=52, 51) | 21.2 [10.1 to 32.3] | 13.7 [4.3 to 23.2]
  Day 337 ACR20 (n=52, 51) | 78.8 [67.7 to 89.9] | 62.7 [49.5 to 76.0]
  Day 337 ACR50 (n=52, 51) | 48.1 [34.5 to 61.7] | 43.1 [29.5 to 56.7]
  Day 337 ACR70 (n=52, 51) | 30.8 [18.2 to 43.3] | 17.6 [7.2 to 28.1]
  Day 421 ACR20 (n=51, 51) | 84.3 [74.3 to 94.3] | 78.4 [67.1 to 89.7]
  Day 421 ACR50 (n=51, 51) | 49.0 [35.3 to 62.7] | 56.9 [43.3 to 70.5]
  Day 421 ACR70 (n=51, 51) | 29.4 [16.9 to 41.9] | 31.4 [18.6 to 44.1]
  Day 505 ACR20 (n=50, 51) | 88.0 [79.0 to 97.0] | 84.3 [74.3 to 94.3]
  Day 505 ACR50 (n=50, 51) | 62.0 [48.5 to 75.5] | 56.9 [43.3 to 70.5]
  Day 505 ACR70 (n=50, 51) | 40.0 [26.4 to 53.6] | 25.5 [13.5 to 37.5]
  Day 561 ACR20 (n=50, 50) | 88.0 [79.0 to 97.0] | 86.0 [76.4 to 95.6]
  Day 561 ACR50 (n=50, 50) | 64.0 [50.7 to 77.3] | 60.0 [46.4 to 73.6]
  Day 561 ACR70 (n=50, 50) | 38.0 [24.5 to 51.5] | 32.0 [19.1 to 44.9]
  Day 645 ACR20 (n=50, 50) | 86.0 [76.4 to 95.6] | 82.0 [71.4 to 92.6]
  Day 645 ACR50 (n=50, 50) | 54.0 [40.2 to 67.8] | 56.0 [42.2 to 69.8]
  Day 645 ACR70 (n=50, 50) | 38.0 [24.5 to 51.5] | 34.0 [20.9 to 47.1]
  Day 729 ACR20 (n=49, 50) | 83.7 [73.3 to 94.0] | 74.0 [61.8 to 86.2]
  Day 729 ACR50 (n=49, 50) | 63.3 [49.8 to 76.8] | 54.0 [40.2 to 67.8]
  Day 729 ACR70 (n=49, 50) | 34.7 [21.4 to 48.0] | 32.0 [19.1 to 44.9]
  Day 813 ACR20 (n=48, 49) | 91.7 [83.8 to 99.5] | 79.6 [68.3 to 90.9]
  Day 813 ACR50 (n=48, 49) | 58.3 [44.4 to 72.3] | 59.2 [45.4 to 72.9]
  Day 813 ACR70 (n=48, 49) | 41.7 [27.7 to 55.6] | 34.7 [21.4 to 48.0]
  Day 897 ACR20 (n=46, 49) | 80.4 [69.0 to 91.9] | 79.6 [68.3 to 90.9]
  Day 897 ACR50 (n=46, 49) | 56.5 [42.2 to 70.8] | 53.1 [39.1 to 67.0]
  Day 897 ACR70 (n=46, 49) | 39.1 [25.0 to 53.2] | 34.7 [21.4 to 48.0]
  Day 981 ACR20 (n=44, 48) | 84.1 [73.3 to 94.9] | 79.2 [67.7 to 90.7]
  Day 981 ACR50 (n=44, 48) | 61.4 [47.0 to 75.8] | 60.4 [46.6 to 74.3]
  Day 981 ACR70 (n=43, 48) | 34.9 [20.6 to 49.1] | 41.7 [27.7 to 55.6]
  Day 1065 ACR20 (n=45, 48) | 80.0 [68.3 to 91.7] | 79.2 [67.7 to 90.7]
  Day 1065 ACR50 (n=45, 48) | 64.4 [50.5 to 78.4] | 60.4 [46.6 to 74.3]
  Day 1065 ACR70 (n=45, 48) | 42.2 [27.8 to 56.7] | 43.8 [29.7 to 57.8]
  Day 1149 ACR20 (n=45, 48) | 84.4 [73.9 to 95.0] | 75.0 [62.8 to 87.2]
  Day 1149 ACR50 (n=45, 48) | 55.6 [41.0 to 70.1] | 62.5 [48.8 to 76.2]
  Day 1149 ACR70 (n=45, 48) | 35.6 [21.6 to 49.5] | 43.8 [29.7 to 57.8]
  Day1233 ACR20 (n=44, 48) | 84.1 [73.3 to 94.9] | 79.2 [67.7 to 90.7]
  Day1233 ACR50 (n=44, 48) | 63.6 [49.4 to 77.9] | 52.1 [38.0 to 66.2]
  Day1233 ACR70 (n=44, 48) | 43.2 [28.5 to 57.8] | 41.7 [27.7 to 55.6]
  Day 1317 ACR20 (n=44, 47) | 90.9 [82.4 to 99.4] | 76.6 [64.5 to 88.7]
  Day 1317 ACR50 (n=44, 47) | 63.6 [49.4 to 77.9] | 53.2 [38.9 to 67.5]
  Day 1317 ACR70 (n=44, 47) | 40.9 [26.4 to 55.4] | 36.2 [22.4 to 49.9]
  Day 1401 ACR20 (n=41, 43) | 90.2 [81.2 to 99.3] | 81.4 [69.8 to 93.0]
  Day 1401 ACR50 (n=41, 43) | 68.3 [54.0 to 82.5] | 51.2 [36.2 to 66.1]
  Day 1401 ACR70 (n=41, 43) | 39.0 [24.1 to 54.0] | 39.5 [24.9 to 54.1]
  Day 1485 ACR20 (n=31, 35) | 83.9 [70.9 to 96.8] | 85.7 [74.1 to 97.3]
  Day 1485 ACR50 (n=31, 35) | 67.7 [51.3 to 84.2] | 62.9 [46.8 to 78.9]
  Day 1485 ACR70 (n=31, 35) | 38.7 [21.6 to 55.9] | 45.7 [29.2 to 62.2]
  Day 1569 ACR20 (n=20, 18) | 100.0 [100.0 to 100.0] | 88.9 [74.4 to 100.0]
  Day 1569 ACR50 (n=20, 18) | 80.0 [62.5 to 97.5] | 72.2 [51.5 to 92.9]
  Day 1569 ACR70 (n=20, 18) | 30.0 [9.9 to 50.1] | 44.4 [21.5 to 67.4]

20. Secondary Outcome: Percentage of Participants With Physical Function Response as Assessed Using the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Improvement is measured by an improved response of at least 0.3 units from baseline on the HAQ-DI score. The HAQ-DI assesses a patient's level of functional ability via 20 questions in 8 categories of functioning. Patients respond on a scale from 0 (no disability) to 3 (completely disabled); total possible score=24. Higher score indicates greater disability. Change from baseline= postbaseline - baseline value.
Time Frame: At Day 1485
Population: All participants who received study drug and who were evaluable
Measure: Number; unit: Percentage of participants
Groups:
- Abatacept, 10 mg/kg: Short-term Period: Participants received a body-weight tiered dose of abatacept approximating 10 mg/kg. Study medication was administered intravenously (IV) on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
- Placebo: Short-term Period: Placebo was administered IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 31 | 35
Percentage of participants | 77.4 | 60.0

21. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI assesses a patient's level of functional ability via 20 questions in 8 categories of functioning. Patients respond on a scale from 0 (no disability) to 3 (completely disabled); total possible score=24. Higher score indicates greater disability. Change from baseline= postbaseline - baseline value.
Time Frame: Day 1485
Population: All participants who received study drug and who were evaluable
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 31 | 35
Units on a scale | -0.76 (0.14) | -0.53 (0.11)

22. Secondary Outcome: Changes From Baseline in Short-Form 36 (SF-36) Physical and Mental Health Summaries
Description: The SF-36 is a 36-item questionnaire used to measure Quality of Life over 8 physically and emotionally based areas: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Answers to each question correspond to a precoded numeric value. An aggregate percentage score is reached for each of the 8 sections and is based on answers to questions. The mean average is worked out for each section. Scores range from 0% (lowest level of functioning) to 100% (highest level of functioning, with higher score indicated increasing levels of functioning.
Time Frame: At Day 1485
Population: All participants who received study drug and who were evaluable
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 31 | 35
Units on a scale
  Physical component score | 10.34 (1.80) | 8.48 (1.57)
  Mental component score | 7.93 (2.44) | 7.73 (2.34)

23. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR)-Defined Low Disease Activity Score (LDAS) and With EULAR-defined Remission
Description: EULAR defines LDAS as a disease activity score as measured by c-reactive protein (DAS28-CRP) ≤3.2 and remission as DAS28-CRP <2.6
Time Frame: At Days 169 and 1485
Population: All participants who received study drug and who were evaluable
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Short-term Period: Participants received placebo IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
Percentage of participants
  EULAR-defined LDAS (Day 169) | 35.8 | 13.5
  EULAR-defined LDAS (Day 1485) (n=31, 35) | 61.3 | 68.6
  EULAR-defined remission (Day 169) | 24.5 | 9.6
  EULAR-defined remission(Day 1485) (n=31, 35) | 35.5 | 54.3

24. Secondary Outcome: Changes From Baseline in the Simplified Disease Activity Index (SDAI) and the Clinical Disease Activity Index (CDAI) Scores
Description: The SDAI is the sum of 5 parameters: Tender joint (TJC) and swollen joint(SJC)counts, based on a 28-joint assessment; patient global (PtGA)and physician global assessments (PGA), assessed on 0-10 cm visual analog scale (VAS), on which higher scores=greater affection due to disease activity DA); and C-reactive protein level. SDAI total score=0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11=low DA, >11 to 26=moderate DA, and >26=high DA. SJC is assessed at each visit, with no swelling=0, swelling=1. TJC is assessed through identification of joints painful under pressure or to passive motion at each visit, with no tenderness=0, tenderness=1. Higher score=greater affection due to DA. CDAI is sum of 4 parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PGA (assessed on 0-10 cm VAS; higher scores=greater affection due to disease activity). CDAI total score=0-76. CDAI <=2.8 indicates disease remission, >2.8 to 10=low DA, >10 to 22=moderate DA, and >22=high DA.
Time Frame: At Days 169 and 1569
Population: All participants who received study drug and who were evaluable
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
Units on a scale
  SDAI score (Day 169) | -22.84 [-26.58 to -19.0] | -14.07 [-17.28 to -10.87]
  SDAI score (Day 1569) (n=20, 18) | -29.74 [-34.06 to -25.43] | -29.20 [-33.70 to -24.70]
  CDAI score (Day 169) | -20.99 [-24.52 to -17.46] | -13.49 [-16.42 to -10.56]
  CDAI score (Day 1569) (n=20, 18) | -27.79 [-31.78 to -23.80] | -27.34 [-31.54 to -23.15]

25. Secondary Outcome: Percentage of Participants With Low Disease Activity Score (LDAS) or Who Are in Remission
Description: LDAS is defined as a Disease Activity Score C-reactive protein (DAS28-CRP) level <=3.2. Remission is defined as a DAS28-CRP level <2.6.
Time Frame: At Days 169, 337, 729, 1149, and 1485
Population: All participants who finished the Short-term period. n=Number of evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Short-term Period: Participants received placebo administered IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
Percentage of participants
  LDAS (Day 169) | 35.8 [22.9 to 48.8] | 13.5 [4.2 to 22.7]
  LDAS (Day 337) (n=52, 51) | 51.9 [38.3 to 65.5] | 35.3 [22.2 to 48.4]
  LDAS (Day 729) (n=48, 50) | 62.5 [48.8 to 76.2] | 56.0 [42.2 to 69.8]
  LDAS (Day 1149) (n=44,48) | 63.6 [49.4 to 77.9] | 60.4 [46.6 to 74.3]
  LDAS (Day 1485) (n=31, 35) | 61.3 [44.1 to 78.4] | 68.6 [53.2 to 84.0]
  Remission (Day 169) | 24.5 [12.9 to 36.1] | 9.6 [1.6 to 17.6]
  Remission (Day 337) (n=52, 51) | 34.6 [21.7 to 47.5] | 23.5 [11.9 to 35.2]
  Remission (Day 729) (n=48, 50) | 43.8 [29.7 to 57.8] | 38.0 [24.5 to 51.5]
  Remission (Day 1149) (n=44,8) | 38.6 [24.2 to 53.0] | 50.0 [35.9 to 64.1]
  Remission (Day 1485) (n=31, 35) | 35.5 [18.6 to 52.3] | 54.3 [37.8 to 70.8]

26. Secondary Outcome: Change From Baseline in Levels of C-reactive Protein (CRP)
Time Frame: Days 169 to 1569
Population: Participants who completed the Short-term Period. n=Number of evaluable participants.
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Placebo: Short-term Period. Participants received placebo IV on Days 1, 15, and 29 and every 28 days thereafter up to and including Day 141. Long-term Period: Participants who completed the Short-term Period received treatment with abatacept, administered IV at a weight-tiered dose approximately 10 mg/kg.
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
mg/dL
  Day 169 | -1.85 (0.29) | -0.58 (0.34)
  Day 197 (n=53, 49) | -1.87 (0.28) | -1.23 (0.36)
  Day 225 | -1.73 (0.51) | -1.62 (0.32)
  Day 253 (n=52, 51) | -1.91 (0.31) | -1.52 (0.32)
  Day 337 (n=52, 51) | -1.94 (0.30) | -1.67 (0.32)
  Day 421 (n=51, 51) | -2.06 (0.26) | -1.77 (0.33)
  Day 505 (n=50, 51) | -2.10 (0.28) | -1.75 (0.33)
  Day 561 (n=50, 50) | -2.23 (0.27) | -1.68 (0.39)
  Day 645 (n=50, 50) | -2.24 (0.28) | -1.88 (0.34)
  Day 729 (n=49, 50) | -2.29 (0.28) | -1.63 (0.37)
  Day 813 (n=48, 49) | -2.24 (0.29) | -1.81 (0.34)
  Day 897 (n=46, 49) | -2.41 (0.30) | -1.76 (0.35)
  Day 981 (n=44, 48) | -1.99 (0.33) | -1.99 (0.36)
  Day 1065 (n=45, 48) | -2.06 (0.32) | -1.47 (0.40)
  Day 1149 (n=45, 48) | -2.00 (0.34) | -1.86 (0.36)
  Day 1233 (n=44, 48) | -1.96 (0.33) | 1.70 (0.37)
  Day 1317 (n=44, 47) | -2.00 (0.35) | -1.81 (0.40)
  Day 1401 (n=41, 43) | -1.93 (0.33) | -1.83 (0.40)
  Day 1485 (n=31, 35) | -1.95 (0.47) | -1.86 (0.41)
  Day 1569 (n=20, 18) | -2.43 (0.43) | -1.68 (0.42)

27. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate
Time Frame: Days 169 to 1569
Population: Participants who completed the Short-term Period. n=Number of evaluable participants.
Measure: Mean (Standard Error); unit: mm/h
Arm/Group | Abatacept, 10 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52
mm/h
  Day 169 | -30.60 (2.93) | -7.12 (3.84)
  Day 197 (n=53, 49) | -28.43 (3.27) | -15.14 (3.79)
  Day 225 | -27.30 (3.09) | -20.27 (3.51)
  Day 253 (n=52, 51) | -27.85 (3.24) | -20.78 (3.97)
  Day 337 (n=52, 51) | -28.58 (3.35) | -23.86 (3.78)
  Day 421 (n=51, 51) | -28.45 (3.34) | -24.94 (3.86)
  Day 505 (n=50, 51) | -31.30 (3.46) | -24.69 (4.07)
  Day 561 (n=50, 49) | -29.32 (3.63) | -24.90 (4.24)
  Day 645 (n=50, 50) | -28.22 (3.74) | -27.38 (4.10)
  Day 729 (n=49, 50) | -32.80 (3.70) | -23.04 (3.60)
  Day 813 (n=48, 47) | -31.52 (3.95) | -22.91 (4.03)
  Day 897 (n=46, 49) | -34.37 (4.13) | -18.22 (4.65)
  Day 981 (n=44, 48) | -33.61 (3.68) | -21.54 (4.53)
  Day 1065 (n=45, 47) | -31.53 (3.95) | -22.09 (4.37)
  Day 1149 (n=45, 48) | -31.00 (4.59) | -20.29 (4.61)
  Day 1233 (n=42, 48) | -30.93 (5.08) | -22.10 (4.70)
  Day 1317 (n=43, 47) | -33.67 (4.45) | -21.89 (4.48)
  Day 1401 (n=41, 43) | -32.41 (4.83) | -23.88 (4.91)
  Day 1485 (n=31, 35) | -33.81 (6.96) | -25.69 (5.70)
  Day 1569 (n=20, 18) | -46.80 (6.79) | -23.33 (5.85)

ADVERSE EVENTS:
Groups:
- Abatacept 10 mg/kg: 500 mg to 1 g; subjects randomized to the abatacept group received a body-weight tiered dose approximating 10 mg/kg. Study medication was administered intravenously (IV) on Days 1, 15, and 29, and every 28 days thereafter up to and including Day 141 (6 month treatment).
Arm/Group | Abatacept 10 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/55 | 3/57
Other Adverse Events (participants affected / at risk) | 27/55 | 26/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 10 mg/kg (N=55) | Placebo (N=57)
ADRENAL CYST (Endocrine disorders) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept 10 mg/kg (N=55) | Placebo (N=57)
WEIGHT INCREASED (Investigations) | 4 | 0
HEADACHE (Nervous system disorders) | 3 | 3
DYSPEPSIA (Gastrointestinal disorders) | 3 | 2
MOUTH ULCERATION (Gastrointestinal disorders) | 3 | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 9
URINARY TRACT INFECTION (Infections and infestations) | 1 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 6
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0
FATIGUE (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.